CLINICAL TRIAL: NCT06701071
Title: Evaluation of a Long Versus Short Clomid Protocol for Controlled Ovarian Stimulation in Patients With Diminished Ovarian Reserve Undergoing In-vitro Fertilization: a Randomized Controlled Trial
Brief Title: Evaluation of a Long Versus Short Clomid Protocol for Controlled Ovarian Stimulation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Richard Paulson, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-23-00039
Record Dates: First submitted 2024-06-13; First posted 2024-11-22 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Clomiphene

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to the two treatment arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Long Clomid (Experimental): Clomid with gonadotropins throughout the entire duration of ovarian stimulation without addition of GnRH antagonist
  Interventions: Drug: Clomiphene Citrate
- 5-day Clomid (Active Comparator): Clomid only for 5 days at beginning of ovarian stimulation with gonadotropins, with GnRH antagonist added when the lead follicle reaches ~14mm.
  Interventions: Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Clomiphene Citrate — Clomiphene citrate is an estrogen receptor antagonist that leads to pituitary FSH release and prevention of the LH surge.

SUMMARY:
The goal of this clinical trial is to evaluate a long Clomid protocol as compared to a 5-day Clomid protocol for ovarian stimulation in patients with diminished ovarian reserve undergoing ovarian stimulation for in-vitro fertilization. The aim of the long Clomid protocol is to intensify stimulation of the ovaries and reduce both cost and injection burden for patients. Participants will be randomized to receive the long Clomid protocol vs. the typical protocol involving Clomid only for 5 days followed by growth hormone-releasing hormone (GnRH) antagonist. The primary outcome the investigators will evaluate will be the number of mature eggs retrieved.

DETAILED DESCRIPTION:
Clomiphene citrate (Clomid) is often used for assisted reproductive technologies and may be used to augment ovarian stimulation with exogenous gonadotropins by stimulating pituitary follicle-stimulating hormone (FSH) release in addition. The mechanism of action of Clomid is antagonism at the estrogen receptor, and this stimulates FSH release from the pituitary. The typical Clomid-based protocol has involved clomid only given for the first five days of stimulation to allow for endometrial development later in the cycle for a fresh embryo transfer following the oocyte retrieval. This protocol involves the addition of a GnRH antagonist medication later in the cycle to prevent premature ovulation. Recent national trends in IVF, however, have moved towards frozen embryo transfers and use of preimplantation genetic testing, which obviates any concerns regarding the endometrium. Recent experience in our clinic has suggested that Clomid may also prevent premature ovulation by antagonizing the positive feedback that is responsible for the luteinizing hormone (LH) surge and ovulation. Given in this manner, Clomid can be given throughout the duration of an ovarian stimulation cycle, achieve higher FSH levels and degree of ovarian stimulation in patients with diminished ovarian reserve, and obviate the need for GnRH antagonist medication (another expensive subcutaneous injection). The objective of this study is to compare a "long Clomid protocol" (i.e. using Clomid throughout the entire duration of the IVF cycle) as compared to the typical 5-day clomid protocol. The investigators hypothesize that the long Clomid protocol will be non-inferior to the typical five-day course and obviate the need for GnRH antagonist by preventing premature ovulation. Patients with diminished ovarian reserve and anticipated poor response to ovarian stimulation will be randomized to the long Clomid protocol vs. a 5-day Clomid with GnRH antagonist protocol. The primary outcome will be oocyte yield. Secondary outcome will be premature ovulation, embryo development, and pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing IVF
* Must meet POSEIDON criteria based on clinic evaluation
* Female partner: Antral follicle count of 2 or more and age <45 at time of stimulation start
* Male partner/sperm source: Cannot be azoospermic
* Planning freeze-all cycle (regardless of blastocyst or cleavage stage culture) or fresh transfer if randomized to short Clomid group
* Planning 36-hour trigger window

Exclusion Criteria:

* Normal ovarian reserve or good response
* Allergy or adverse reaction to Clomid
* Minimal stimulation protocols
* History of prior premature ovulation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females can undergo ovarian stimulation
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of mature oocytes | Up to 1 month after study completion
  The number of mature oocytes retrieved at oocyte retrieval

SECONDARY OUTCOMES:
Number of participants that experience premature ovulation | Up to 1 month after study completion
  Premature LH surge, progesterone rise and estradiol decrease, or evidence of premature ovulation (no oocytes on retrieval or free fluid and follicular collapse on ultrasound)
Number of oocytes that get fertilized and grow to the blastocyst stage | Up to 1 month after study completion
  Fertilization rate and blastulation
Pregnancy outcomes | Up to 3 years after study completion
  Clinical pregnancy rate, ongoing pregnancy rate, live birth rate

CONTACTS AND LOCATIONS:
Overall Officials: Richard Paulson, Principal Investigator — paulsonivf@havingbabies.com
Locations (1):
- HRC Fertility, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No